CLINICAL TRIAL: NCT02311959
Title: Therapeutic Nipple Areola Skin-sparing Mastectomy.
Brief Title: Therapeutic Nipple Sparing Mastectomy.
Acronym: MAPAM-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14 SEIN 10
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Breast; Invasive carcinoma; In situ carcinoma; Mastectomy; Nipple areola; Reconstruction; Local recurrence
MeSH Terms: conditions — Breast Neoplasms; Carcinoma in Situ | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Invasive or in situ breast carcinoma. (Experimental)
  Interventions: Procedure: Nipple sparing mastectomy

INTERVENTIONS:
Procedure: Nipple sparing mastectomy — Standardized surgical procedure by :
  * Nipple sparing mastectomy with nipple core histopathology.
  * Immediate breast reconstruction (flap and/or implant).
  * +/- lymph node evaluation (sentinel node procedure or axillary dissection).

SUMMARY:
This is a phase III, multicentric, single arm study with a sequential design using the exact conditional Poisson test.

The primary objective of this prospective study is to evaluate whether selected breast carcinoma patients could be treated with nipple sparing mastectomy (NSM) with an acceptable low local recurrence rates.

450 patients will be included over a period of 4 years and will be followed for a 5 years period (twice a year).

All patients must have a complete preoperative evaluation (bilateral mammography, bilateral breast ultrasonography +/- MRI), and a histopathological diagnostic proof of carcinoma (invasive or in situ, all histopathological types, first treatment or relapse).

The study procedure is represented by nipple areola skin-sparing mastectomy followed by immediate breast reconstruction.

After surgery, early and late complications, including specific complications (suffering of the nipple-areolar complexe and suffering of the skin flaps), will be evaluate.

An esthetic evaluation (by patient and clinician) and a quality of life evaluation will be realized throughout the study.

A complementary study, prospective, non-interventional, will be proposed to patients who will benefit from the same surgical technique (NSM) followed by immediate reconstruction, but in the context of preventive surgery (prophylactic surgery for patients mutated or high genetic risk). The aim of this complementary study, which will include a maximum of 60 patients, is to evaluate associated morbidity in prophylactic NSM.

Data will be collected over a 3 months period after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with invasive breast carcinoma stage T1 or T2 and / or in situ (any histological type) proved on histopathological diagnosis.
* Patient with an indication of total mastectomy.
* Patient without preoperative indication of adjuvant radiotherapy according to regional and / or national guidelines.
* Disease located more than 2 cm from the nipple after complete clinical and radiologic breast evaluation (mammography, ultrasound +/- MRI).
* Initial breast cancer or recurrence.
* Patient wishing to receive immediate breast reconstruction.
* WHO performance < or = 2.
* Patient older than 40 years.
* For patients of childbearing age, use an effective contraceptive methods for the duration of the study.
* For patients of childbearing potential, negative pregnancy test available before inclusion.
* Patient affiliated to a social health insurance in France.
* Patient who signed informed consent before enrollment in the study and before any specific procedure for the study.

Exclusion Criteria :

* Positive node on physical examination or proved by cytology.
* Combination of 2 predictive factors of postoperative radiotherapy : macroscopic multifocal, grade 2 or 3, vascular emboli, overexpressed HER2 (human epidermal growth factor receptor-2), triple negative (Estrogen Receptor, Progesterone Receptor and HER2 negative).
* Neoadjuvant treatment for the current disease.
* Patient with bilateral breast cancer.
* Paget disease.
* T3 or T4 carcinoma.
* Metastatic breast cancer (disease staging realized according to national or regional guidelines).
* Breast hypertrophy requiring a nipple support flap.
* Nursing or pregnant woman.
* Patient participating in any other interventional clinical study.
* Any psychological, familial, geographic or social situation not to comply with medical monitoring and/or procedures in the study protocol.
* Patient protected by law.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Local recurrence rate. | 9 years.
  Annual incidence of local recurrence defined by the number of local recurrences (skin, thoracic wall and nipple) among the patient years of follow-up..

SECONDARY OUTCOMES:
Early and late complications | 9 years.
  Early and late complications will be evaluated using NCI toxicity scale version 4.0.
Disease free Survival. | 9 years.
  Disease-free survival is the period between the date of origin and date of the first event as defined below, or date of latest news (Censored Data).
  The events included in the definition of disease-free survival are local recurrence, lymph node metastases, contralateral locations, distant metastases, second breast cancer and death from any causes.
Metastasis Free Survival. | 9 years.
  Metastasis free survival is defined as the time from inclusion until the date of metastasis recurrence or the date of the latest news (Censored data).
Overall Survival. | 9 years
  Overall survival is defined as the time from inclusion until the date of death or the date of the latest news (Censored data).
Aesthetic evaluation. | 9 years.
  The aesthetic evaluation will be realized by both the surgeon and the patient using to the Licket scale.
Quality of life. | 9 years.
  The quality of life will be evaluated according to the Breast-Q questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eva JOUVE, Md., Principal Investigator — IUCT-O
Locations (33):
- France (33):
  - Centre Hospitalier de Blois, Blois
  - Institut Bergonie, Bordeaux
  - Pôle santé Léonard de Vinci, Chambray-lès-Tours
  - Centre Georges Francois Leclerc, Dijon
  - Hôpital privé Drôme Ardèche, Guilherand-Granges
  - Clinique du Mail, La Rochelle
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Clinique Saint Amé, Lambres-lez-Douai
  - Hopital de Levallois-Perret, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Institut Paoli Calmettes, Marseille
  - Clinique Clementville, Montpellier
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Institut Du Cancer de Montpellier, Montpellier
  - Centre Antoine LACASSAGNE, Nice
  - Hôpital Européen Georges Pompidou, Assistance Publique - Hôpitaux de Paris, Paris
  - Ap-Hp - Hopital Tenon, Paris
  - CHRU Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Mathilde, Rouen
  - Hôpital René Huguenin, Saint-Cloud
  - Clinique Mutualiste Chirurgicale, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne
  - Etablissement Rennais du Sein - CHP St Grégoire, Saint-Grégoire
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Clinique Saint Jean, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Filleron T, Lusque A, Dalenc F, Ferron G, Roche H, Martinez A, Jouve E. Alternative methodological approach to randomized trial for surgical procedures routinely used. Contemp Clin Trials. 2018 May;68:109-115. doi: 10.1016/j.cct.2018.03.016. Epub 2018 Mar 30. PMID 29608972